CLINICAL TRIAL: NCT06571513
Title: Written Exposure Therapy to Improve Recovery Among Sexual Assault Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-1437
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Trauma and Stressor Related Disorders; Mental Disorders; Stress Disorders, Traumatic; Stress Disorders, Post-traumatic; Sexual Assault
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Trauma and Stressor Related Disorders; Mental Disorders; Stress Disorders, Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written Exposure Therapy (Experimental): Five sessions of remotely-delivered written exposure therapy.
  Interventions: Behavioral: Written Exposure Therapy
- Unemotional Writing (Placebo Comparator): Five sessions of remotely-delivered non-emotional writing.
  Interventions: Behavioral: Unemotional Writing

INTERVENTIONS:
Behavioral: Written Exposure Therapy — During session one of the written exposure therapy intervention, the therapist will provide psychoeducation about PTSD and the rationale for the proposed intervention. Psychoeducation and treatment rationale are scripted to ensure consistency. The therapist will provide the participant with instructions for writing about the same trauma memory (their recent sexual assault) during each session. They will be asked to look back at the event and write for 30 minutes about the details of the event including what they saw, heard, felt, smelled, etc. without regard for spelling or grammar. The participant will self-report Subjective Units of Distress Scale (SUDS) levels to the therapist at the beginning and end of each session. After 30 minutes, the therapist will ask the participant to stop writing, review the experience of writing and discuss as needed, and conclude the session.
  Arms: Written Exposure Therapy
Behavioral: Unemotional Writing — During the unemotional writing sessions, the therapist will read instructions for writing about non-emotional topics. The participant will be instructed to describe what they did the day before the session from the time they woke up until the time they went to bed, as objectively as possible, without regard for spelling or grammar. The therapist will then leave the participant with a written version of the instructions for 30 minutes while the participant writes. The participant will self report Subjective Units of Distress Scale (SUDS) levels to the therapist at the beginning and end of each session. After 30 minutes, the therapist will ask the participant to stop writing, review the experience of writing and discuss as needed, and conclude the session.
  Arms: Unemotional Writing

SUMMARY:
The main objective of this pilot trial is to determine the feasibility and initial efficacy of telehealth-delivered written exposure therapy to reduce the development of posttraumatic stress disorder after sexual assault. This pilot trial will provide the data necessary to design and support a large-scale trial.

DETAILED DESCRIPTION:
Each year, approximately 100,000 women in the United States present to sexual assault nurse examiner (SANE) programs for evaluation after experiencing sexual assault. A wealth of data demonstrates that the development of adverse posttraumatic neuropsychiatric sequelae such as posttraumatic stress disorder (PTSD) is common in this population and that individuals with a history of traumatic stress exposure and/or posttraumatic stress symptoms are at increased risk. Unfortunately, no secondary preventive interventions are currently widely available that can prevent PTSD among those at high risk. Moreover, the 10% of sexual assault survivors in the United States who live in rural communities face even greater barriers to obtaining care. Written exposure therapy is an evidence-based, low-cost intervention that has demonstrated efficacy in treating chronic PTSD symptoms after a variety of traumatic stress exposures, including sexual assault. In addition, telehealth delivery of written exposure therapy for PTSD has yielded similar treatment outcomes and lower attrition compared to in-person delivery. The present protocol will assess the feasibility and preliminary efficacy of telehealth-delivered written exposure therapy as a secondary preventive intervention for sexual assault survivors in the acute aftermath of trauma exposure. This pilot trial will randomize N=80 women who received SANE care following sexual assault to five sessions of either virtual written exposure therapy (n=40) or virtual unemotional writing control (n=40). The same experienced therapists will deliver both interventions via telehealth/video sessions. Participant follow-ups will be performed remotely via REDCap self-report surveys by trained assessors and research associates. Results of this trial will demonstrate the feasibility and potential efficacy of written exposure therapy to reduce the development of PTSD after sexual assault and will provide the data necessary to design and support a large-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender woman
* Writes and speaks English
* 18+ years of age
* Presents for SANE care within 7 days of sexual assault
* Discharged home after SANE care
* Has an email address
* Has an Apple (iOS) or Android-compatible smartphone with photo capability (for writing session upload), without loss of cellular connection due to inability to pay bill for >1 year
* Willing to participate in remote therapy sessions
* Meets PTSD risk score criteria
* Meets with research assistant (RA) for informed consent within 30 days of SANE care

Exclusion Criteria:

* Age <18
* Pregnant
* Incarcerated or in police custody
* Presented for SANE care >7 days after assault
* Has had a change in psychiatric medication regimen 1 month prior to study enrollment
* Currently receiving cognitive-behavioral therapy or exposure-based psychological treatment
* Sexually assaulted at work or by a colleague
* Currently lives with the person who assaulted them
* History or condition that in investigator's judgment would likely make a participant non-compliant/unsuitable for participation, including deafness or blindness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifies as a woman
Enrollment: 80 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Changes in PTSD Symptom Severity Over Time | Baseline, Week 4, Week 8, Month 3, Month 5
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure designed to assess PTSD symptoms as defined by the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5). Each item of the PCL-5 is scored on a five-point scale ranging from 0 ("not at all") to 4 ("extremely"). Items are summed to provide a total severity score (range = 0-80), with higher scores indicating greater symptom severity. PTSD symptom severity will be compared between treatment groups over time.
Recruitment Rates | Baseline
  To assess feasibility of the study recruitment protocol, the proportion of eligible participants who enroll in the study and are randomized will be calculated.
Retention Rates | Month 5
  To assess feasibility of the study protocol, the proportion of participants who complete the study protocol, according to study arm and in total, will be calculated.
Treatment Completion Rates | Week 8
  To assess feasibility of the treatment protocol, treatment completion rates will be calculated according to study arm and in total. Treatment completers will be defined as participants who complete at least 4 out of 5 written exposure therapy or control sessions.

SECONDARY OUTCOMES:
Change in Pain Symptom Severity and Extent Over Time | Baseline, Week 4, Week 8, Month 3, Month 5
  Pain severity and extent will be evaluated using a modified version of the Regional Pain Scale, where each item is scored on a 0-10 numeric rating with 0 indicating no pain and 10 indicating severe pain. Pain symptom severity and extent will be compared between treatment groups over time.
Change in Somatic Symptom Score Over Time | Baseline, Week 4, Week 8, Month 3, Month 5
  Somatic symptoms will be assessed using a modified version of the Pennebaker Inventory of Limbic Languidness (PILL), which assesses the frequency of common physical symptoms and sensations. Each item is scored on a 0-10 scale where 0 indicates no problems. Number of moderate to severe somatic symptoms (scores ≥ 4) will be compared between groups.
Change in Depressive Symptom Score Over Time | Baseline, Week 4, Week 8, Month 3, Month 5
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form 8b is an 8-item scale developed to assess depression in individuals 18 and older. Each item is rated on a five-point scale. For this study, response options are slightly altered for greater consistency across measures and precision in response levels (i.e., 1 = "never" is changed to none of the time and 5 = "always" is changed to "all or almost all of the time."). Items are summed to provide a total severity score (range = 8-40), with higher scores indicating greater severity of depression. Depressive symptom severity will be compared between treatment groups over time.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A McLean, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared on request provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Time Frame: Beginning 12 months following publication and continuing for 36 months
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.